CLINICAL TRIAL: NCT02114918
Title: Attention Training for Childhood Obsessive Compulsive Disorder
Acronym: AMP-OCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Susanna Chang, PhD, Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB#11-000195; 1R34MH095885-01A1 (NIH)
Record Dates: First submitted 2014-04-11; First posted 2014-04-15 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Obsessive Compulsive Disorder
Keywords: obsessive compulsive disorder; children; adolescents; attention bias modification
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Adenosine Monophosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Attention Modification Program (Experimental): Active computer-based attention training treatment designed to directly but implicitly modify biased attention patterns in anxious patients in service of symptom relief. AMP is a modified version of the dot-probe paradigm similar to the original task used by MacLeod, Mathews, and Tata. This paradigm has been modified to facilitate an attention bias away from threatening material. In this case, the probe always replaces the neutral word.
  Interventions: Behavioral: Attention Modification Program
- Attention Control Condition (Placebo Comparator): Control computer-based attention training task, which is not designed to modify biased attention patterns in anxious patients. ACC is a modified version of the dot-probe paradigm similar to the original task used by MacLeod, Mathews, and Tata. In this case, the probe randomly replaces the neutral word or the threat word.
  Interventions: Behavioral: Attention Control Condition

INTERVENTIONS:
Behavioral: Attention Modification Program — Each trial begins with a fixation cross presented in the center of the computer screen for 500 ms. The cross is then replaced by a word pair presented in the center of the screen for 500 ms. The word pair disappears and a probe (i.e., the letter "E" or "F") appears immediately in the location of one of the two words. Participants will be instructed to decide whether the letter is an E or an F and press the corresponding mouse button. This paradigm has been modified to facilitate an attention bias away from threatening material. In this case, the probe always replaces the neutral word. Thus, although there will be no specific instruction to direct attention away from the threat word, on all trials, the position of the neutral word will indicate the position of the probe.
  Other Names: AMP, attention bias modification, attention training
  Arms: Attention Modification Program
Behavioral: Attention Control Condition — Each trial begins with a fixation cross presented in the center of the computer screen for 500 ms. The cross is then replaced by a word pair presented in the center of the screen for 500 ms. The word pair disappears and a probe (i.e., the letter "E" or "F") appears immediately in the location of one of the two words. Participants will be instructed to decide whether the letter is an E or an F and press the corresponding mouse button. This paradigm is not intended to facilitate an attention bias away from threatening material. In this case, the probe randomly replaces the threat or neutral word.
  Other Names: ACC
  Arms: Attention Control Condition

SUMMARY:
Voluntary and involuntary attention processes are thought to play an important role in the development and maintenance of anxiety disorders including OCD. Individuals with OCD pay greater attention to threat information related to their illness and have difficulty shifting their attention from such triggers. Studies suggest that a change in attention bias may lead to a change in anxiety vulnerability. However, few studies have directly examined the causal role of attention bias in the maintenance of anxiety underlying OCD and whether modification of such biases may reduce pathological anxiety symptoms particularly in children. In this proposal, we aim to translate basic findings from research on cognitive biases in anxiety into a novel computerized intervention for child Obsessive Compulsive Disorder (OCD). The treatment is designed to target a basic cognitive vulnerability in OCD, namely the selective processing of threatening OCD-related information. 52 children with OCD will be randomly assigned to either a 12-session attention modification program (AMP) or an attention control condition (ACC). Clinical assessment of symptom severity along with a brief neurocognitive battery will be conducted before and after treatment. We hypothesize that children in the AMP group at end of treatment will show (1) decreased attention bias to OCD-related triggers using an independent measure of attention bias to assess change and (b) reduced OCD severity. This study is an initial step towards demonstrating the feasibility and efficacy of a novel computerized attention training program for OCD that ultimately may prove to be a highly transportable and accessible intervention for this childhood psychiatric disorder. Furthermore, the project will also examine neurocognitive performance before and after attention training to elucidate possible predictors and mechanisms of treatment response.

DETAILED DESCRIPTION:
In this proposal, we aim to translate basic findings from research on cognitive biases in anxiety into a novel computerized intervention for child OCD. The treatment is designed to target a basic cognitive vulnerability in OCD, namely the selective processing of threatening OCD-related information. Briefly, the computerized procedure involves repeatedly redirecting participants' attention away from OCD-relevant threat cues in order to induce selective processing of neutral (non-threat) stimuli. This study is an initial step towards demonstrating the efficacy of a potentially highly transportable and accessible intervention for OCD. Furthermore, the project will also examine neurocognitive performance before and after attention modification to elucidate possible predictors and mechanisms of treatment response.

Aim 1: To examine the preliminary efficacy of a 12-session computerized attention modification program (AMP) on attention bias and symptom severity in children with OCD.

Hypothesis 1a: AMP treatment compared to the attention control condition (ACC) will be associated with a decrease in attention bias towards threat-cues in youth with OCD.

Hypothesis 1b: AMP treatment will be associated with a decrease in OCD symptom severity among OCD youth as measured by clinician-administered diagnostic interview and symptom rating scales.

Aim 2: To examine the changes in neurocognitive status over the course of treatment with AMP in children and adolescents with OCD.

Hypothesis 2: Those children who respond to AMP will exhibit improved performance on relevant neurocognitive measures at post-treatment.

Aim 3: To examine the relationship between baseline neurocognitive status and response to AMP.

Hypothesis 3: Baseline neurocognitive performance will be associated with greater AMP-related improvement in symptom severity among youth with OCD.

Exploratory Aim: To investigate the potential relationship between AMP and changes in behavioral and electrophysiological (EEG) correlates of cognitive control and affect regulation before and after treatment with AMP or ACC. The objective is to examine the feasibility, acceptability and suitability of using Error-Related Negativity (ERN), an evoked response potential (ERP) generated from cognitive activation paradigms assessing action-monitoring and conflict resolution under neutral and emotional contexts, to elucidate potential neural mechanisms underlying treatment. Although not powered for formal tests of mediation, we will explore in a preliminary fashion whether these neural indices may serve as potential biomarkers for pediatric OCD as well as predictors/mediators of treatment response.

Preliminary hypotheses: 1) Youth with OCD will be characterized by high amplitude ERN, which will not change with treatment; 2) AMP treatment will be associated with changes in EEG reflecting greater engagement of top-down (as indexed by the P3 component) versus bottom-up (indexed by the P1/N1 components) neural processes, particularly among children who exhibit improved performance on cognitive control tasks; 3) Baseline executive functioning in interference control and action monitoring will be associated with greater AMP-related improvement in OCD severity; 4) We will also explore the relationships of key variables such as trait anxiety, self-reported attention control, baseline OCD symptom severity and attention bias with each other and with response to AMP.

OCD is a chronic and often disabling psychiatric condition, affecting 2-4% of children and adolescents1. In the absence of effective treatment, it is often associated with considerable social, academic and familial impairment along with considerable psychiatric comorbidity including Tourette's and other Chronic Tic Disorders. Although a number of empirically supported treatments, both behavioral and pharmacological, exist for OCD, many children and their families are either not able to adequately access these treatments or derive only partial benefit from them. Thus, it is of critical importance to expand treatment options and develop more effective treatments that have the potential to be widely accessible to children suffering from OCD.

One etiological model of OCD proposes that symptoms arise from the abnormal processing of threat-relevant information. According to this model, selective attention to threatening information heightens anxiety and anxiety-related avoidance of the perceived threat, and the avoidance behaviors, in turn, prevent disconfirmation of fear-related beliefs and serves to maintain anxiety. Thus, attention bias towards threat may be causally related to the behavioral avoidance of the perceived threat. Research indicates that attention bias towards OCD related material ameliorates after effective cognitive behavioral therapy, thus highlighting that attention bias is malleable. Nevertheless, the critical question remains whether a reduction in attention bias causes a reduction in OCD symptoms or whether attention bias is an epiphenomenon of the symptoms. Recently, studies have begun to directly manipulate attention bias to address this question. In one such study, attention was trained in adults with OCD contamination fears by building a contingency between the locations of the OCD-related word in the active condition and not in the control condition on a modified dot-probe task. Participants in the attention training group showed significant reductions in both attention bias for threat and OCD symptom severity. The extension of this research to clinical patient and child samples with a multi-session treatment protocol has yet to be conducted. To date, no study has investigated attention training in children with OCD, although there are data to suggest positive results in adults with OCD as well as Social Phobia and Generalized Anxiety Disorder.

A number of recent studies have demonstrated that the willful direction of attention in the presence of threatening stimuli activates prefrontal regions thought to be involved in attention control, which in turn appears to down-regulate activation of the amygdala, a structure involved in the emotional processing of fear/threat stimuli. Many of these tasks have involved techniques like cognitive reappraisal or altering cognitive processing of threatening. The question remains whether similar neurobiological mechanisms underlie the effects of attention training. Given the importance of higher-level attention control in reducing biased attention processing and dampening anxious states, helping anxious individuals improve attention control may be an important mechanism for reducing the negative impact and development of psychopathology. In an attempt to gather preliminary data on the possible neurocognitive predictors and mechanisms of treatment response, we also plan to assess aspects of response inhibition and memory/learning that have been implicated in neurocognitive studies of OCD before and after treatment with AMP.

We hypothesize that training attention away from OCD-related threat stimuli will decrease attention bias towards the threat and based on the assumption that attention bias is causally related to anxiety symptoms, this decrease in bias would lead to a decrease in avoidance of threatening stimuli. More specifically, we predict that compared to the control condition (ACC), AMP will decrease attention bias towards the threat and facilitate behavioral approach towards the feared stimuli in children with OCD along with an overall decrease in their symptom severity.

The present study focuses on children and adolescents for two important reasons. First, OCD typically onsets in childhood, and enhanced understanding of the neuro-developmental correlates of OCD and mechanisms underlying treatment at this age has the potential to prevent long-term morbidity. Second, the focus on this age group allows us to study the disorders prior to the development of significant secondary psychiatric and psychosocial morbidity, which commonly accompanies OCD in adulthood. Thus far, only limited research on the effects of attention modification training on OCD severity has been conducted in children. This study may generate significant new information concerning the neurocognitive underpinnings of OCD, the commonality of these underpinnings to other neurodevelopmental disorders of childhood, and the neurocognitive correlates of response to a potentially new and relatively accessible nonpharmacological treatment intervention. This knowledge will be used to develop more effective treatments with an eye towards matching interventions to specific individuals on the basis of characteristic pre-treatment cognitive profiles.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-17 (inclusive) at the time of initial evaluation
* Subject meets Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) diagnostic criteria for OCD.
* Unmedicated or on stable medication treatment for anxiety, OCD, attention deficit hyperactivity disorder, tics, and/or depressive disorder for at least 6 weeks prior to study entry, with no planned changes for duration of study participation.
* Child is fluent English speaker.
* Parental informed consent and child informed assent must be completed. Parents must agree to their child's participation in this protocol.

Exclusion Criteria:

* Intelligence Quotient < 80 on Wechsler Abbreviated Scale of Intelligence (WASI).
* Excessive or problematic substance use as reported per initial telephone screening, or DSM-IV Conduct Disorder within the past 3 months.
* Subject has a lifetime DSM-IV diagnosis of pervasive developmental disorder, Mania, or Psychotic Disorder.
* Subject has any serious psychiatric, psychosocial, or neurological condition (i.e., attention deficit hyperactivity disorder, major depressive disorder, anxiety, anxiety, severe aggression, family discord) requiring immediate treatment other than that provided in the current study.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2013-04; Primary Completion 2016-01 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression-Severity (CGI-S) and Improvement (CGI-I) Scales Change From Pre-Treatment to Post-Treatment | pre-treatment (week 0) and post-treatment (week 5)
  Clinical Global Impression-Severity (CGI-S) and Improvement (CGI-I) Scales. The CGI-S and CGI-I are clinician-rated scales used in clinical trials for over 25 years. Participants receiving a post-treatment CGI-I score of 1 (very much improved) or 2 (much improved) on this one-item, 7-point rating will be considered treatment responders.

SECONDARY OUTCOMES:
Children's Yale-Brown Obsessive Compulsive Scale Change From Pre-Treatment to Post-Treatment | pre-treatment (week 0) and post-treatment (week 5)
  Children's Yale Brown Obsessive Compulsive Scale (CYBOCS) is a psychometrically sound, semi-structured clinical interview assessing OCD severity. The measure includes a comprehensive symptom checklist and will be used as one measure of treatment response.
Attention Bias Assessment Change from Pre-Treatment to Post-Treatment | pre-treatment (week 0) and post-treatment (week 5)
  Computerized assessment of attention bias. The classic dot-probe paradigm used in the majority of studies examining attention bias will be adapted for this project. AMP will occur with one set of words (e.g., Set A) and the other word set (Set B) will be used for pre and post-training assessment of attention bias. We plan to use a modified version of the Posner spatial cueing paradigm using 8 OCD-related threat and eight neutral word cues word pairs.

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Chang, PhD, Principal Investigator — University of California, Los Angeles; John Piacentini, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Semel Institute for Neuroscience and Human Behavior, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No